CLINICAL TRIAL: NCT06384807
Title: A Phase 1/2, First in Human, Dose Escalation and Dose Expansion Study of BHV-1510 (Previously PBI-410) as Monotherapy and in Combination With Anti-Cancer Agents in Participants With Advanced Solid Tumors
Brief Title: A Phase 1/2 Study of BHV-1510 (Previously PBI-410) in Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biohaven Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Organization: Biohaven Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BHV1510-101 (PBI-410-101)
Record Dates: First submitted 2024-04-22; First posted 2024-04-25 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumor
Keywords: Trop2 targeting ADC; Antibody-drug conjugate; Trop2; ADC
MeSH Terms: interventions — cemiplimab

STUDY DESIGN:
Intervention Model Description: Dose escalation followed by enrollment in signal-finding cohorts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BHV-1510 Monotherapy Dose Escalation (Experimental)
  Interventions: Drug: BHV-1510
- BHV-1510 in combination with Cemiplimab dose escalation (Experimental)
  Interventions: Drug: BHV-1510; Drug: Cemiplimab

INTERVENTIONS:
Drug: BHV-1510 — BHV-1510 will be administered on Day 1 every 3 weeks
  Other Names: PBI-410; GQ1010
Drug: Cemiplimab — cemiplimab (350mg) will be administered as an IV infusion on Day 1 every 3 weeks
  Arms: BHV-1510 in combination with Cemiplimab dose escalation
Drug: BHV-1510 — BHV-1510 will be administered on Day 1 every 2 weeks
  Other Names: PBI-410; GQ1010
Drug: BHV-1510 — BHV-1510 will be administered on Day 1 and Day 8 every 3 weeks
  Other Names: PBI-410; GQ1010
Drug: Cemiplimab — cemiplimab (350mg) will be administered as an IV infusion on Day 1 and Day 8 every 3 weeks
  Arms: BHV-1510 in combination with Cemiplimab dose escalation

SUMMARY:
This is a Phase 1/2, first in human (FIH), open-label, multicenter study of BHV-1510 monotherapy and in Combination with Cemiplimab in participants with previously treated, advanced solid tumors.

DETAILED DESCRIPTION:
This is a Phase 1/2, first in human (FIH), open-label, multicenter study of BHV-1510, a Trop-2 directed antibody-drug conjugate (ADC), in participants with previously treated, advanced solid tumors. The study comprises 2 parts: a Phase 1 Dose Escalation and a Phase 2 Dose Expansion. The Phase 1 will investigate the safety and tolerability of BHV-1510 given in monotherapy and given in combination with cemiplimab and identify one or more recommended doses for expansion (RDEs) and the maximum-tolerated dose (MTD) (if one exists). Once the RDE has been established, Phase 2 will open to investigate the preliminary efficacy of BHV-1510 in signal-finding expansion cohorts.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female participants aged ≥18 years.
* Unresectable, incurable, locally advanced or metastatic epithelial-origin solid tumor that is refractory to standard therapies, or has no approved standard therapies, or no approved standard therapies at its current treatment stage. If applicable to the tumor type, participants must have received platinum-based chemotherapy, standard of care immunotherapy, and standard of care targeted therapies.
* Measurable disease (per RECIST 1.1).
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1.
* Participants have adequate hematologic, renal, liver, and coagulation function as defined by the following (blood transfusion or growth factor support is not allowed within 7 days prior to blood samples that will be used to establish eligibility):

  * Hemoglobin ≥9 g/dL
  * Absolute neutrophil count >1,500/mm3; participants with known Duffy null phenotype who have absolute neutrophil count ≥1,200/mm3 may be enrolled
  * Platelets >100,000/mm3
  * Creatinine clearance ≥50 mL/min measured or estimated using the Cockcroft-Gault formula; 24-hour urine collection is allowed, but not required.
  * Total bilirubin ≤1.5 × upper limit of normal (ULN); participants with known Gilbert's syndrome who have total bilirubin level ≤3×ULN may be enrolled.
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <2.5×ULN (or ≤5×ULN for participants with hepatic metastases)
  * Alkaline phosphatase <2.5×ULN (or ≤5×ULN for participants with hepatic and/or bone metastases)
  * International normalized ratio (INR) or prothrombin time (PT) ≤1.5×ULN
  * Activated partial thromboplastin time (aPTT) ≤1.5×ULN. Study participants on therapeutic doses of anticoagulation medication must have INR and/or aPTT ≤ the upper limit of the therapeutic range for intended use
* Have recovered (ie, improvement to Grade 1 or better) from all acute toxicities from previous therapy, excluding alopecia and vitiligo.

BHV-1510 in Combination with specific inclusion criteria:

* histologically or cytologically documented advanced (locally, recurrent, inoperable, cannot be treated with curative intent) or metastatic cancer.
* received ≤ 2 prior lines of systemic anti-cancer therapy and at most one prior anti-programmed cell death protein 1 (PD-1) (programmed death-ligand 1 [PD-L1]) therapy for advanced/ metastatic disease.

Key Exclusion Criteria:

* Women who are pregnant or lactating.
* Clinically significant intercurrent disease.
* Has symptomatic brain metastases or has had any radiation or surgery for brain metastases within 4 weeks of C1D1.
* Has clinically significant corneal disease.
* Requires supplemental oxygen for daily activities.
* Previous treatment with a Trop-2-targeted therapy, including Trop-2 ADCs.
* Has a medical history of interstitial lung disease (eg, noninfectious interstitial pneumonia requiring steroid treatment, pneumonitis, pulmonary fibrosis, or severe radiation pneumonitis) or current interstitial lung disease or are suspected to have any of these diseases based on imaging at Screening.
* Any standard cancer therapy (eg, chemotherapy, hormonal therapy, radiotherapy, immunotherapy, biologic therapy treatment) or experimental therapy within 3 weeks or 5 half-lives, whichever is shorter, prior to C1D1. The interval may be reduced to 2 weeks for bone and visceral metastasis therapy. Any major surgical procedure within 6 weeks prior to C1D1.
* History of severe hypersensitivity reactions to other monoclonal antibodies or either the drug substances or inactive ingredients of BHV-1510.
* Has current or previously treated leptomeningeal carcinomatosis.
* Use of OAP1B1 and OATP1B3 inhibitors within 14 days prior to starting trial.

BHV-1510 in Combination Specific Exclusion Criteria:

* Hypersensitivity to cemiplimab or any of its excipients or contraindicated to cemiplimab per approved local labeling.
* Experienced Grade 3 or higher immune-related AEs with prior treatment of anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX 40, CD137).
* Prior allogeneic stem cell or solid organ transplantation.
* Patients with history of myocarditis.
* Presence of cardiovascular disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Number of patients with adverse events (AEs) | Through study completion, estimated as an average of 47 months
  Description: Incidence and severity of AEs, serious adverse events (SAEs) and dose limiting toxicities (DLTs). Severity of AEs will be assessed according to the NCI CTCAE v5.0. This applies to both the BHV-1510 monotherapy arm and BHV-1510 in combination with Cemiplimab arm.
Phase 1: Recommended doses or schedules for expansion (RDEs) and maximum tolerated dose (MTD) | Approximately 15 months
  Based on tolerability and preliminary antitumor activity. This applies to both the BHV-1510 monotherapy arm and BHV-1510 in combination with Cemiplimab arm.
Phase 2: Objective Response Rate (ORR) for BHV-1510 for monotherapy and in combination with cemiplimab | Through study completion, estimated as an average of 47 months
  Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1.
Phase 2: Number of patients with AEs for BHV-1510 for monotherapy and in combination with cemiplimab | Through study completion, estimated as an average of 47 months
  Incidence and severity of AEs, SAEs and DLTs. Severity of AEs will be assessed according to the NCI CTCAE v5.0
Phase 2: Duration of Response (DoR) for BHV-1510 for monotherapy and in combination with cemiplimab | Through study completion, estimated as an average of 47 months
  Assessed by RECIST v 1.1

SECONDARY OUTCOMES:
Phase 1 and 2: Maximum Plasma Concentration (Cmax) of BHV-1510, total antibody and payload (BHC-0080269) | Up to 8 timepoints, but not exceeding, 22 days in Cycles 1 and 3
Phase 1 and 2: Area Under the Concentration versus time Curve from the end of infusion to the last measurable concentration (AUClast) of BHV-1510, total antibody and payload | Up to 8 timepoints, but not exceeding, 22 days in Cycles 1 and 3
Phase 1 and 2: Area Under the Concentration versus time curve extrapolated to infinity (AUCinf) of BHV-1510, total antibody and payload | Up to 8 timepoints, but not exceeding, 22 days in Cycle 1
Phase 1 and 2: Area under the concentration versus time curve over the dosing interval (AUCtau) of BHV-1510, total antibody and payload | Up to 8 timepoints, but not exceeding, 22 days in Cycles 1 and 3
Phase 1 and 2: Elimination half-life (t1/2) of BHV-1510, total antibody and payload | Up to 8 timepoints, but not exceeding, 22 days in Cycles 1 and 3
Phase 1 and 2: Trough concentration (Ctrough) of BHV-1510, total antibody and payload | Up to 8 timepoints, but not exceeding, 22 days in Cycles 1 and 3
Phase 1 and 2: Total body clearance (CL) after IV administration or apparent total body clearance (CL/F) after SC administration of BHV-1510 and total antibody | Up to 8 timepoints, but not exceeding, 22 days in Cycles 1 and 3
Phase 1 and 2: Percent bioavailability (%F) after SC administration of BHV-1510 and total antibody | Up to 8 timepoints, but not exceeding, 22 days in Cycles 1 and 3
Phase 1 and 2: Volume of distribution at steady state (Vss) after IV administration or apparent volume of distribution at steady state (Vss/F) after SC administration of BHV-1510 and total antibody | Up to 8 timepoints, but not exceeding, 22 days in Cycles 1 and 3
Phase 1: ORR | Through study completion, estimated as an average of 47 months
  Assessed by RECIST v 1.1. This applies to both the BHV-1510 monotherapy arm and BHV-1510 in combination with Cemiplimab arm.
Phase 1: Duration of Response (DoR) | Through study completion, estimated as an average of 47 months
  Assessed by RECIST v 1.1. This applies to both the BHV-1510 monotherapy arm and BHV-1510 in combination with Cemiplimab arm.
Phase 1 and 2: Immunogenicity of BHV-1510 | Through study completion, estimated as an average of 47 months
  Incidence of ADA at baseline and post-treatment, including ADA titer
Phase 2: Disease control rate (DCR) for BHV-1510 for monotherapy and in combination with cemiplimab | Through study completion, estimated as an average of 47 months
  Assessed by RECIST v 1.1
Phase 2: Progression free survival (PFS) for BHV-1510 for monotherapy and in combination with cemiplimab | Through study completion, estimated as an average of 47 months
  Assessed by RECIST v 1.1
Phase 2: Overall survival (OS) for BHV-1510 for monotherapy and in combination with cemiplimab | Through study completion, estimated as an average of 47 months
  OS is defined as the time period from the start of administration to death due to any cause
Phase 2: Effects of BHV-1510 monotherapy and payload on the QTc interval using the Fridericia's correction method (QTcF), and on other ECG parameters (heart rate [HR], PR, and QRS interval) | Approximately 15 months

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Biohaven Pharmaceuticals, Inc.
Locations (17):
- United States (17):
  - Site-113, Duarte, California
  - Site-112, La Jolla, California
  - Site-111, Palo Alto, California
  - Site-114, Washington D.C., District of Columbia
  - Site-103, Miami, Florida
  - Site-105, Orlando, Florida
  - Site-115, Tampa, Florida
  - Site-110, Augusta, Georgia
  - Site-109, Detroit, Michigan
  - Site-101, St Louis, Missouri
  - Site-117, New York, New York
  - Site-116, Oklahoma City, Oklahoma
  - Site-108, Philadelphia, Pennsylvania
  - Site-107, Nashville, Tennessee
  - Site-104, Dallas, Texas
  - Site-106, West Valley City, Utah
  - Site-102, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No